CLINICAL TRIAL: NCT03898232
Title: A Single Surgeon Retrospective Cohort Study of Clinical and Radiological Outcomes Among Patients Treated With Lumbar Interbody Fusion Augmented With Prosidyan Fibergraft® Putty for Degenerative Spinal Disease
Brief Title: Fibergraft Interbody Fusion Retrospective
Acronym: FIFR
Status: Completed | Type: Observational
Sponsor: Bone and Joint Clinic of Baton Rouge (Other)
Responsible Party: Sponsor
Other Study IDs: FIFR-28
Record Dates: First submitted 2019-03-20; First posted 2019-04-01 (Actual); Last update posted 2021-01-29 (Actual); Status verified 2021-01

CONDITIONS: Degenerative Disc Disease; Degenerative Spondylolisthesis; Spinal Degeneration; Spinal Stenosis
MeSH Terms: conditions — Intervertebral Disc Degeneration; Spinal Stenosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Device: Yes

INTERVENTIONS:
Radiation: Computed Tomography (CT) Scan of the Lumbar Spine — Patients in the cohort who have not received a 12 month post-op CT scan will be asked to enroll in the study and undergo a CT of the lumbar spine.

SUMMARY:
A single center study of clinical and radiological outcomes in a retrospective cohort of patients treated with Lumbar Interbody Fusion augmented with Prosidyan Fibergraft for 1 or 2 level degenerative spinal disease by a single surgeon.

Study Design: Retrospective chart review with prospective data collection.

DETAILED DESCRIPTION:
Background and Rationale: Degenerative pathologies of the lumbar spine including degenerative disc disease, spondylosis and spondylolisthesis are the leading indications for lumbar interbody fusion (LIF) among low back pain patients. Prosidyan's Fibergraft is a bioactive synthetic bone graft substitute that is ultraporous and made from bioactive glass fibers. The proposed study will be an analysis of clinical outcomes among patients who underwent lumbar interbody fusion augmented with Prosidyan Fibergraft by a single surgeon.

Objective(s):

PRIMARY: To assess the fusion rate in this retrospective cohort at 12 months post-operatively.

SECONDARY:

* To report and analyze trends (if any) among diagnosis, number of levels, approach (TLIF, LIF or ALIF) and fusion status.
* To assess pain and functional health changes pre to post-operatively. SAFTEY: To report the rate of surgical adverse events and subsequent surgeries at the operative level.

Study design: Retrospective chart review with prospective data collection.

Procedures: Patients will be screened by retrospective chart review. Eligible patients will be contacted and asked to participate. Consenting patients will answer questionnaires and undergo a CT lumbar scan.

Study Product / Intervention: The device under investigation is Prosidyan Fibergraft. However, since study subjects are retrospectively enrolled, they will have received the device before entering the study.

ELIGIBILITY:
Inclusion Criteria:

* - Previous Lumbar Interbody Fusion (LIF) at 1-3 levels augmented with Prosidyan Fibergraft Putty.
* No revision or device removal at the operative level(s).
* Patient did not undergo a Lumbar CT at least 8 months post-operatively.
* Willing and able to sign Informed Consent.
* Willing and able to complete questionnaires and undergo CT scan of the Lumbar Spine

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who underwent a Lumbar Interbody Fusion (LIF) at 1-3 levels augmented with Prosidyan Fibergraft Putty.
Sampling Method: Non-Probability Sample
Enrollment: 66 (Actual)
Dates: Start 2019-05-09 (Actual); Primary Completion 2020-02-20 (Actual); Study Completion 2020-02-20 (Actual)

PRIMARY OUTCOMES:
Fusion Rate | 12 months post-operatively
  The primary outcome for this study will be the overall fusion rate in the retrospective cohort. Fusion will be assessed from a Lumbar CT scan. The criteria used to assess fusion status will be according to the scale developed by Brantigan, Steffee, and Fraser (BSF criteria).

SECONDARY OUTCOMES:
Mean change in Visual Analog (VAS) Pain scale | Pre-operatively to 12 months post-operatively
  Mean change in low back pain as measured by a 100 mm Visual Analog Scale where 0 indicates no pain and 100 indicates the greatest pain.
Mean change in Oswestry Disability Index (Function) score | Pre-operatively to 12 months post-operatively
  Mean change in low back functional status as measured by the Oswestry Disability Index where a score of 0 indicates no disability and a score of 100 represents maximum disability

CONTACTS AND LOCATIONS:
Locations (1):
- Bone and Joint Clinic of Baton Rouge, Baton Rouge, Louisiana, United States